CLINICAL TRIAL: NCT03205319
Title: To Scope or Not to Scope: Trial to Reduce Inappropriate Oesophagogastroduodenoscopies for Dyspepsia; a Randomised Controlled Trial
Brief Title: Trial to Reduce Inappropriate Oesophagogastroduodenoscopies for Dyspepsia
Acronym: TRIODe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Maastricht University Medical Center (Other); Canisius-Wilhelmina Hospital (Other); VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-3079; NL.60056.091.17 (Other: ToetsingOnline)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2018-10

CONDITIONS: Dyspepsia; Indigestion
Keywords: Oesophagoduodenoscopy; E-learning; Appropriate use of healthcare; Deimplementation
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: Multicenter, randomised controlled, open label
Masking Description: Masking will be impossible in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm / e-learning (Experimental): Patients will receive e-learning instead of upper GI endoscopy.
  Interventions: Device: e-learning
- Control arm / upper GI endoscopy (No Intervention): Patients will receive the upper GI endoscopy, i.e. standard of care

INTERVENTIONS:
Device: e-learning — The e-learning for patients is a user friendly, audiovisual based, online-accessible program, designed especially for this study. The e-learning will contain information on dyspepsia and advice on lifestyle interventions
  Arms: Intervention arm / e-learning

SUMMARY:
Indigestion or dyspepsia is highly prevalent worldwide. Often these symptoms are of benign nature and subside without treatment, or with lifestyle interventions like dietary modifications. Too often, gastroscopy is performed because of dyspepsia. Although this is indicated when malignancy is suspected, in a substantial part of the cases the gastroscopy is not indicated and will not achieve clinically relevant results. It is suspected that gastroscopy is often used for reassurance of patients or as a 'last resort'.

Our hypothesis is that adequate education of patients can replace this need for invasive measures. The aim of this study was therefore to reduce the volume of gastroscopies for dyspepsia, by offering patients an e-learning containing educational material on dyspepsia.

During the trial, 119 dyspeptic patients, referred for gastroscopy by the GP, will randomly be divided into two groups: One group will receive the e-learning instead of gastroscopy (intervention), the other group will receive the gastroscopy (control).

After a twelve week follow-up, change in symptom severity, disease specific quality of life and fear of disease will be compared between the two groups.

DETAILED DESCRIPTION:
Rationale: Upper gastrointestinal (GI) symptoms, such as dyspepsia without alarm symptoms, are highly prevalent in the general population. Lifestyle modifications and medication can reduce symptoms in most patients. Guidelines state that oesophagogastroduodenoscopy (OGD) is only indicated in a selected high risk group. In spite of these guidelines, OGD referrals for dyspepsia without alarm symptoms are still substantial, subjecting patients to unnecessary risks and causing a burden on healthcare costs and endoscopic capacity. Therefore a strategy is needed to reduce the volume of OGDs in dyspepsia without alarm symptoms.

Objective: To evaluate the clinical use of a patient-centred, education based, clinical strategy to reduce the volume of endoscopies for dyspepsia in patients over 18 years of age without alarm symptoms, referred for OGD through open-access endoscopy compared to usual care.

Study design: A multicentre, randomised, controlled superiority trial, with two parallel arms and a primary endpoint of the percentage of patients receiving OGD. Intervention and usual care will be compared.

Study population: 119 Patients, aged 18 years or above, with upper GI symptoms without alarm symptoms, referred for open-access OGD.

Intervention: Patients will be offered e-learning instead of endoscopy. The e-learning will contain educational material and questionnaires. Questionnaire data will be extracted from the e-learning.

Main study endpoints: The main study endpoint is the difference in proportion of patients receiving OGD between both arms and Patient Reported Outcomes (PROMS), after a follow-up of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Reported upper gastrointestinal symptoms in the past 6 months
* Referred for OGD
* Guidelines for referral not met
* Signed informed consent

Exclusion Criteria:

Patients who fulfil the criteria for OGD according to the Dutch college of General Practitioners (NHG) guidelines and NICE guidelines on 'Upper gastrointestinal tract cancers'.

In addition, patients with:

* A family history of gastric- or oesophageal cancer (at least one first or second grade family member with a malignancy at the age of 50 or younger)
* Diseases or circumstances that will most likely impair understanding of the e-learning
* Any argument provided by a patient's own GP stating the urge of OGD, notwithstanding the guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
The difference in proportion performed OGDs between groups | 12 weeks
  The difference between the two study arms in proportion of patients that have received OGD, measured 12 weeks after the initial visit to the endoscopy clinic, out of the total number of patients referred for open-access endoscopy

SECONDARY OUTCOMES:
The influence of the intervention on health-related anxiety | 12 weeks
  The difference between the change scores of the two study arms concerning health-related anxiety, measured by the total score on the validated Short Health Anxiety Inventory
The influence of the intervention on severity of upper GI symptoms | 12 weeks
  The difference between the change scores of the two study arms concerning severity of upper GI symptoms, measured by the mean on the subscale scores of the validated PAGI-SYM questionnaire
The influence of the intervention on dyspepsia-related quality of life | 12 weeks
  The difference between the change scores of the two study arms concerning dyspepsia-related quality of life, measured by the sum of the subscale scores of the validated Nepean Dyspepsia Index
The ability of the e-learning to improve knowledge | 15 minutes
  Using a knowledge test integrated in the e-learning and administered before and after the e-learning, the difference in correctly answered questions will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Drenth, MD, PhD, Principal Investigator — Radboud University Medical Center; Prof. Dr. Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (5):
- Netherlands (5):
  - Ziekenhuis Gelderse Vallei, Ede, Gelderland
  - Canisius-Wilhelmina Hospital, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - VieCuri Medical Center, Venlo, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Jong JJ, Lantinga MA, Tan ACITL, Aquarius M, Scheffer RCH, Uil JJ, de Reuver PR, Keszthelyi D, Westert GP, Masclee AAM, Drenth JPH. Web-Based Educational Intervention for Patients With Uninvestigated Dyspepsia Referred for Upper Gastrointestinal Tract Endoscopy: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jun 1;181(6):825-833. doi: 10.1001/jamainternmed.2021.1408. PMID 33900373